CLINICAL TRIAL: NCT01374009
Title: H1N1 Vaccine in Pregnancy: a Registry for the Fall and Winter of 2009
Status: Terminated | Type: Observational
Why Stopped: Participants were consented but registry was not developed due to low numbers
Sponsor: Dalhousie University (Other)
Collaborators: Li Ka Shing Foundation (Other); PHAC/CIHR Influenza Research Network (Other Government)
Responsible Party: Principal Investigator, Shelly A. McNeil, MD, Dalhousie University
Other Study IDs: 114141
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Vaccine Exposure During Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study it to rapidly create a brief registry of pregnant women who receive the H1N1 vaccine in Ontario, British Columbia, and Nova Scotia during the pandemic H1N1 2009/2010 influenza season.

DETAILED DESCRIPTION:
For Part 1, a brief amount of data will be collected on each woman at the time of her vaccination. These data will be filled out on a single data collection sheet by her Obstetrics Clinic physician or nurse, which will be completed at the time of her vaccination.

For Part 2, after a woman's expected delivery date, data sources will be used for participants. Two groups of non-vaccinated controls will be derived from the provincial perinatal databases:

1. The active non-vaccinated controls will be recruited from the concurrent year, matched to women who were vaccinated in 2009/2010. For each of the three perinatal databases, 5 non-vaccinated active controls will be matched by maternal age +/- 3 years, same-hospital delivery, and delivery date +/- 7 days.
2. The passive non-vaccinated controls will be derived from the preceding year (i.e., 2008). For each of the three perinatal databases, 5 non-vaccinated passive controls will be matched by maternal age +/- 3 years, same-hospital delivery, and delivery date +/- 7 days.

For women who delivered in Ontario, the Niday Perinatal Database will be used. (https://www.nidaydatabase.com/info/index.shtml).

For women who deliver in British Columbia, their data will be linked to the British Columbia Perinatal Database Registry (http://www.bcphp.ca/Database%20Content.htm). Women who deliver in Nova Scotia will be linked to Nova Scotia Atlee Perinatal Database (http://rcp.nshealth.ca/rcp_3347.html).

Information that will be obtained is as follows:

* Actual delivery date (DD/MM/YYYY)
* Number of infants delivered
* Mode of delivery (vaginal for Caesarean)
* Liveborn or stillborn
* Presence of a congenital anomaly
* Presence of intrauterine growth restriction or small-for-gestational age birthweight
* Presence of a neonatal infection
* Presence of neonatal sepsis
* Need for ventilation of the neonate
* Need for Neonatal Intensive Care of the Neonate.

For Part 3, between 18-24 months after a woman's actual delivery date, a woman may be telephoned at her home to ask her about the health and developmental milestones of her baby. This phase may or may not be done, but consent will be obtained nonetheless.

ELIGIBILITY:
Inclusion Criteria:

* Received the H1N1 vaccine during pregnancy

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who recieved the H1N1 vaccine during pregnancy in 2009.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelly A McNeil, MD FRCPC, Principal Investigator — Queen Elizabeth II Health Sciences Centre, Dalhousie University, Halifax, NS; Joel Ray, MD FRCPC, Principal Investigator — St. Michael's Hospital/University of Toronto, Toronto, Ontario; Alison McGeer, MD MSc FRCPC, Principal Investigator — Mount Sinai Hospital/University of Toronto, Toronto, Ontario; Deborah Money, MD FRCSC, Principal Investigator — University of British Columbia, Vancouver, British Columbia; Graeme N Smith, MD PhD FRCSC, Principal Investigator — Queen's Inversity, Kingston, Ontario; Jennifer Blake, MD MSc FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre and Women's College Hospital, University of Toronto; Mark Yudin, MD MSc FRCSC, Principal Investigator — St. Michael's Hospital, University of Toronto, Toronto, Ontario; Muhammad Mamdani, PharmD MPH, Principal Investigator — Li Ka Shing Knowledge Institute, St. Michael's Hospital, University of Toronto, Toronto, Ontario
Locations (7):
- Canada (7):
  - Children's and Women's Health Centre, University of British Columbia, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Queen's University, Kingston, Ontario
  - Li Ka Shing Knoweldge Institute, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre and Women's College Hospital, Toronto, Ontario